CLINICAL TRIAL: NCT05171218
Title: The Effects of Music & Auditory Beat Stimulation on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Lucid, Inc. (Industry); Mitacs (Industry)
Responsible Party: Principal Investigator, Frank Russo, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 2020-068
Record Dates: First submitted 2021-11-27; First posted 2021-12-28 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Anxiety
Keywords: Anxiety; Auditory Beat Stimulation; Binaural Beats; Mental Health; Music; Neuroscience; Psychology
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Participants taking anxiolytics (n = 163) were randomly assigned to a single 24- minute session of sound-based treatment: combined (Music with theta auditory beat stimulation), music-alone, theta auditory beat stimulation-alone, or pink noise (control). Pre- and post-intervention somatic and cognitive state anxiety measures (STICSA State) were collected along with trait anxiety (STICSA Trait), personality measures (Short Form Eysenck Personality Inventory) and musical preferences (Short Test of Music Preferences).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Music & Auditory Beat Stimulation (Experimental): Participants listened to calm music with theta auditory beat stimulation for 24 minutes
  Interventions: Behavioral: Music & Auditory Beat Stimulation
- Music Alone (Active Comparator): Participants listened to calm music for 24 minutes
  Interventions: Behavioral: Music Alone
- Auditory Beat Stimulation (Active Comparator): Participants listened to theta auditory beat stimulation for 24 minutes
  Interventions: Behavioral: Auditory Beat Stimulation
- Pink Noise (Sham Comparator): Participants listened to pink noise for 24 minutes
  Interventions: Behavioral: Pink Noise

INTERVENTIONS:
Behavioral: Music & Auditory Beat Stimulation — Listening to calm music and auditory beat stimulation Participants listened to calm music with theta auditory beat stimulation for 24 minutes
  Arms: Music & Auditory Beat Stimulation
Behavioral: Music Alone — Listening to calm music Participants listened to calm music for 24 minutes
  Arms: Music Alone
Behavioral: Auditory Beat Stimulation — Listening to theta auditory beat stimulation Participants listened to theta auditory beat stimulation for 24 minutes
  Arms: Auditory Beat Stimulation
Behavioral: Pink Noise — Listening to pink noise Participants listened to pink noise for 24 minutes
  Arms: Pink Noise

SUMMARY:
Anxiety is a growing problem and has been steadily increasing, particularly in the adolescent and young adult populations in the past 24 years. Music and auditory beat stimulation (ABS) in the theta frequency range (4-7 Hz) are sound-based anxiety treatments that have been independently investigated in prior studies. Here, the anxiety-reducing potential of calm music combined with theta ABS was examined in a large sample of participants. Participants taking anxiolytics (n = 163) were randomly assigned to a single 24-minute session of sound-based treatment: combined (music & ABS), music-alone, ABS-alone, or pink noise (control). Pre- and post-intervention somatic and cognitive state anxiety measures (STICSA State) were collected along with trait anxiety (STICSA Trait), personality measures (Short Form Eysenck Personality Inventory) and musical preferences (Short Test of Music Preferences).

DETAILED DESCRIPTION:
In this study, the investigators examined and compared the effectiveness of ABS in the theta range, calm music playlist curated by an affective music recommendation system, and the combination of ABS and the same music to reduce anxiety and stress levels (as measured by the State Trait Inventory for Cognitive and Somatic Anxiety (STICSA)) compared to a control condition (pink noise). Prior work has demonstrated that ABS and music both reduce anxiety when presented on their own. It is hypothesized that music with ABS will lead to significantly lower anxiety levels and increased calmness compared to the other experimental conditions. Approximately 163 participants were recruited from the Prolific online participant pool (https://www.prolific.co). The experiment was conducted on the Qualtrics survey platform, and the experimental treatment was provided with the LUCID Research App. After reading and agreeing with the consent form, participants provided their Prolific ID and then filled out the Short Test of Music Preferences (STOMP), Queen's Music Questionnaire, Anxiety coping method's questionnaire, Positive and Negative Affect Scale (PANAS), Self-Assessment Manikin (SAM), Eysenck Personality Questionnaire, and the State Trait Inventory of Cognitive and Somatic Anxiety (STICSA). Participants were also asked to list any medications currently being taken (including cannabis). Participants were then randomly assigned to one of four treatment groups: (1) music; (2) music and auditory beat stimulation (ABS); (3) auditory beat stimulation (ABS) alone; or (4) pink noise for 24 minutes. Participants then received instructions on how to download the LUCID Research app on their iOS device or access the LUCID Research App through a virtual machine using their computer. Participants listened to their randomly assigned treatment for 24 minutes. Participants then completed their post-intervention questionnaires which included: the STICSA state version, SAM and PANAS. The investigators' hypotheses were that the combined, music alone and ABS alone conditions would experience a greater reduction in somatic and cognitive state anxiety compared to the pink noise control condition. These hypotheses were pre-registered using the Open Science Framework (Registration DOI: https://doi.org/10.17605/OSF.IO/VHCA5) and were based upon previous studies showing that ABS and music listening are capable of reducing anxiety. The investigators had no specific predictions for moderate and high trait anxiety participants, but their pre-registration noted their intention to recruit from both of these populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+)
* Must be taking anxiety medication
* Self-identified normal hearing
* No known cardiac issues
* No known epilepsy/seizures

  * Have access to an iOS device (iPhone or iPad) to run the Research Application

Exclusion Criteria:

* Adults younger than 18
* Not taking anxiety medication
* Have known cardiac issues

  - Do not have access to an iOS device (iPhone or iPad) to run the Research Application
* Have known epilepsy/seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Anxiety: State Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | 24 minutes
  The State Trait Anxiety Inventory for Cognitive and Somatic Anxiety has good reliability and validity as a measure of state and trait cognitive and somatic anxiety. The minimum score is 10 and the maximum is 40. Higher scores indicate higher anxiety (worse outcome). But in this study the post-intervention anxiety score is subtracted from the pre-intervention anxiety score, giving a measure of anxiety reduction. In the case of this anxiety reduction measure, higher anxiety reduction scores would indicate a better outcome.

SECONDARY OUTCOMES:
Mood: Positive and Negative Affect Scale (PANAS) | 24 minutes
  The Positive and Negative Affect Scale has good reliability and validity and has been widely used in many studies to assess mood. This scale generates two scores: 1) Positive affect (higher score indicates a better outcome), scores range from 10-50. 2) Negative affect (higher score indicates worse outcome), scores range from 10-50.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Russo, PhD, Study Director — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We have registered the project on Open Science Framework and will make all elements of IPD open to the public. Please see: https://osf.io/efya2/ Study protocol and analysis plan: https://doi.org/10.17605/ OSF.IO/VHCA5 Consent form: https://osf.io/efya2/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are available now and will be for 7 years post data collection completion as per our REB approval: approximately January 2028
Access Criteria: There is no specific access criteria for the IPD on OSF. It is freely and openly available to anyone.
URL: https://osf.io/efya2/

REFERENCES:
- [Background] Bados A, Gomez-Benito J, Balaguer G. The state-trait anxiety inventory, trait version: does it really measure anxiety? J Pers Assess. 2010 Nov;92(6):560-7. doi: 10.1080/00223891.2010.513295. PMID 20954057
- [Background] Gray EK, Watson, D. Assessing positive and negative affect via self-report. In: Coan JA, Allen, J.J.B., editor. Handbook of emotion elicitation and assessment. New York, NY: Oxford University Press; 2007.
- [Background] Gros DF, Antony MM, Simms LJ, McCabe RE. Psychometric properties of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA): comparison to the State-Trait Anxiety Inventory (STAI). Psychol Assess. 2007 Dec;19(4):369-81. doi: 10.1037/1040-3590.19.4.369. PMID 18085930
- [Background] Phillips SP, Yu J. Is anxiety/depression increasing among 5-25 year-olds? A cross-sectional prevalence study in Ontario, Canada, 1997-2017. J Affect Disord. 2021 Mar 1;282:141-146. doi: 10.1016/j.jad.2020.12.178. Epub 2020 Dec 30. PMID 33418360
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Davis WB, Thaut MH. The Influence of Preferred Relaxing Music on Measures of State Anxiety, Relaxation, and Physiological Responses. Journal of Music Therapy. 1989;26(4):168-87. doi: 10.1093/jmt/26.4.168.
- [Background] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Background] McConnell PA, Froeliger B, Garland EL, Ives JC, Sforzo GA. Auditory driving of the autonomic nervous system: Listening to theta-frequency binaural beats post-exercise increases parasympathetic activation and sympathetic withdrawal. Front Psychol. 2014 Nov 14;5:1248. doi: 10.3389/fpsyg.2014.01248. eCollection 2014. PMID 25452734
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Background] Wahbeh H, Calabrese C, Zwickey H. Binaural beat technology in humans: a pilot study to assess psychologic and physiologic effects. J Altern Complement Med. 2007 Jan-Feb;13(1):25-32. doi: 10.1089/acm.2006.6196. PMID 17309374
- [Background] Yusim A, Grigaitis J. Efficacy of Binaural Beat Meditation Technology for Treating Anxiety Symptoms: A Pilot Study. J Nerv Ment Dis. 2020 Feb;208(2):155-160. doi: 10.1097/NMD.0000000000001070. PMID 31977827
- [Background] Bringman H, Giesecke K, Thorne A, Bringman S. Relaxing music as pre-medication before surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2009 Jul;53(6):759-64. doi: 10.1111/j.1399-6576.2009.01969.x. Epub 2009 Apr 14. PMID 19388893
- Available data/document: Individual Participant Data Set — https://osf.io/efya2/
- Available data/document: Study Protocol — https://doi.org/10.17605/OSF.IO/VHCA5
- Available data/document: Statistical Analysis Plan — https://doi.org/10.17605/OSF.IO/VHCA5
- Available data/document: Informed Consent Form — https://osf.io/efya2/

DOCUMENTS (3):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05171218/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05171218/SAP_001.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05171218/ICF_002.pdf